# Gentle Warriors Academy Healthy Marriage and Responsible Fatherhood Program Evaluation

4/22/2024

Clinicaltrials.gov ID: NCT06899100

**Study Protocol** 

# PROGRAM BACKGROUND

#### 1. PROGRAM SUMMARY

Please provide a brief summary of your grant project including the needs to be addressed, the services provided, and the population served.

Gentle Warriors Academy (GWA) is designed to help urban community adult fathers age 18 and older with dependent child(ren) up to 24 years of age incorporate practices and behaviors for managing the responsibilities of being parents/co-parents and partners through responsible parting, healthy marriage/relationships, economic stability activities, and grant-funded participation supports through a 40-hr/10-week cohort-based approach. These core areas are reinforced through GWA's coordinated case management process and wrap-around services, which is tailored to help address obstacles that fathers and their families face on their journeys to attaining and maintaining healthy parental and partner relationships as well as program completion.

Fathers Incorporated utilizes a skills-based curricula for its core GWA services: Next Level Fatherhood which was created and tailored by subject matter experts and Fathers Incorporated practitioners/staff to address the complex challenges and needs of urban community fathers. All curricula consist of 10 modules of learning that are designed to develop practical and comprehensive skillsets that are transferrable throughout all aspects of life.

The objectives of the Next Level Fatherhood curriculum are to: 1. Provide participants with practical skills necessary to navigate critical aspects of responsible fatherhood, healthy marriages, and personal/family economic stability; 2. Provide participants with tools that will assist them in strengthening their marriages, child engagement, and co-parenting relationships, and to provide information and resources around viable economic stability for themselves and their families; 3. Provide participants with skills necessary to making better and more informed parenting choices, to be more pro-active and less reactive, and to strengthen parental relationships; and 4. Encourage participants to become more acutely aware of how they present themselves in the lives of their children, significant others, an in the "systems" (family court, judicial court, child support, state agencies etc.) in which they have to navigate.

Participating fathers will work with Case Managers to review the results of all assessments and to determine necessary support services through the duration of program participation. Case Managers will implement case management best practices, record case notes that document interaction/support provided to all participants and will ensure that each participant receives six hours of dedicated case management from program enrollment through completion. Certified Life Coaches will work in tandem with Case Managers to help participants obtain and reach their goals, promote, and develop their strengths, and to overcome difficult challenges, specifically within their marriages or other significant relationships, their economic viability and their parental responsibilities as identified through co-developed Individual Success Plans (ISPs).

#### 2. EVALUATION GOALS

Please briefly describe key goals of your evaluation and what you hope to learn below.

In this evaluation, it is anticipated that participants will show an increase in:

- Communications and handling conflict and other related relationship skills
- Understanding in role as a father
- Improved communication with partner/co-partner
- Understanding the quality of father-child engagement
- Various forms of contact with children

# 3. EVALUATION ENROLLMENT

Please provide the expected start and end dates for program and evaluation enrollment using the tables below. For impact studies, please indicate expected start and end dates for each study group.

| DESCRIPTIVE EVALUATION Please leave blank if not conducting a descriptive outcome evaluation. | | |
|---|---|---|
| | Program Enrollment Study Enrollment | |
| Start Date | 4/1/2021 | 4/1/2021 |
| End Date | 7/1/2025 | 3/31/2024 |
| Definition | All program participants who enroll in services | All program participants who consent to being part of the study |

# 4. EVALUATION TIMELINE

Please include a timeline for key activities of the evaluation below. Example of activities may include IRB submission, staff training, waves of data collection, analysis period, and report writing and submission.

| Evaluation Activity | Start Date | End Date |
|---|---|---|
| Additional Evaluation staff hiring and onboarding | 1/15/2021 | 2/15/2021 |
| Evaluation staff training | 1/22/2021 | 2/20/2021 |
| Evaluation Kickoff meeting and orientation with all program staff | 2/2/2021 | 2/3/2021 |
| IRB training and certification by all program and evaluation staff | 10/1/2020 | 2/28/2021 |
| Development and submission of Evaluation Plan document | 1/15/2021 | 2/19/2021 |
| Evaluation Tools Development | 10/1/2021 | 2/28/2021 |
| IRB Approval | 3/1/2021 | 3/15/2021 |
| IRB Full Board Approval | 05/11/2023 | 06/01/2024 |
| IRB Approval for Incarcerated Population | 06/02/2023 | 06/01/2024 |
| CQI Team Formed and Meeting bi-weekly | 3/15/2021 | 7/1/2025 |
| Training for CQI Team | 3/15/2021 | 3/28/2021 |
| Training for all Program Staff on Research Methods and process | 3/15/2021 | 3/28/2021 |
| Implementation Evaluation Data Collection | 4/1/2021 | 8/15/2025 |
| -Baseline | 4/1/2021 | 7/1/2025 |
| -Post Test | 5/15/2021 | 8/15/2025 |
| -Follow-up | 4/1/2021 | 8/15/2025 |
| 1 <sup>st</sup> Manuscript submitted for publication | 7/1/2025 | 9/30/2025 |

# **EVALUATION PLAN**

#### 1. RESEARCH QUESTIONS

#### 1.1. OVERVIEW OF RESEARCH QUESTIONS

Please state the research questions(s) that the evaluation intends to answer and for each research question indicate the type: implementation or outcome.

- o Implementation Questions: Identifying whether a program has been successful in attaining desired implementation goals (e.g., reaching intended target population, enrolling intended number of participants, delivering training and services in manner intended, etc.)
- Outcome Questions: Identifying whether program is associated with intended outcomes for participants (e.g., do participants' knowledge, attitudes, behaviors, or awareness change?)

Research questions in this study are framed by a Descriptive Evaluation Design to assess whether outcomes improve for low-income fathers who participate in the Gentle Warriors Academy (GWA) Project. Primary outcomes are assessed before and after participants complete core curricula—Next Level Fatherhood—and Case Management and Certified Life Coaching as support services (pre to post). Primary outcomes will indicate whether behavior improved for healthy family relationships (parent, co-parent, and partner). See Table 1 below.

| No | Research Question | Implementation or Outcome? |
|---|---|---|
| R1 | Will participants report significantly <b>healthier parenting behavior</b> after completing primary educational services and employment support services? | Primary Outcome |
| R2 | Will participants report significantly <b>healthier parenting attitudes</b> after completing primary educational services and employment support services? | Primary Outcome |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

| R3 | Will participants report significantly <b>healthier co-parenting behavior</b> after completing primary educational services and employment support services? | Primary Outcome |
|---|---|---|
| R4 | Will participants report significantly <b>healthier partner relationship behavior</b> after completing primary educational services and employment support services? | Primary Outcome |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 1.2. OUTCOME RESEARCH QUESTIONS

For each <u>outcome research question</u> listed above, whether a descriptive or impact design, summarize the inputs (e.g., program components, program supports, implementation features, etc.), target population (e.g., the population for which the effect will be estimated) and the outcomes (e.g., child well-being, father-child engagement, etc.) that will be examined to answer the research question(s). Comparisons for descriptive evaluations may reflect circumstances before the grant, pre-treatment, or pre-determined benchmark from other studies with similar interventions.

| Research<br>Question<br>Number<br>Should<br>correspond<br>to the<br>number<br>indicated<br>in Table<br>1.1 above | Intervention Program component or set of activities that the evaluation will test or examine | Target Population Population for which the effect of the treatment will be estimated | Comparison What the intervention will be compared to (e.g., pre-intervention for descriptive designs) | Outcome Changes that are expected to occur as a result of the intervention | Confirmatory or Exploratory? Confirmatory: those upon which conclusions will be drawn Exploratory: those that may provide additional suggestive evidence |
|---|---|---|---|---|---|
| R1 | Primary curricula (Next Level Fatherhood); Support Services (Case Management, Life Coaching); | Urban fathers<br>who are 18+<br>years with<br>children up to<br>24 years | Assessment of healthy parenting behavior at GWA Project enrollment. | Participants who complete primary and support services will report healthier parenting behavior | Confirmatory |

| | Continuous<br>Quality<br>Improvement<br>(CQI) Process | | | one year<br>after GWA<br>Project<br>enrollment. | |
|---|---|---|---|---|---|
| R2 | Primary curricula (Next Level Fatherhood); Support Services (Case Management, Life Coaching); Continuous Quality Improvement (CQI) Process | Urban fathers<br>who are 18+<br>years with<br>children up to<br>24 years | Assessment of healthy parenting attitudes at GWA Project enrollment. | Participants who complete primary and support services will report healthier parenting attitudes one year after GWA Project enrollment. | Confirmatory |
| R3 | Primary curricula (Next Level Fatherhood); Support Services (Case Management, Life Coaching); Continuous Quality Improvement (CQI) Process | Urban fathers<br>who are 18+<br>years with<br>children up to<br>24 years | Assessment of healthy coparenting behavior at GWA Project enrollment. | Participants who complete primary and support services will report healthier coparenting behavior one year after GWA Project enrollment. | Confirmatory |
| R4 | Primary curricula (Next Level Fatherhood); Support Services (Case Management, Life Coaching); Continuous Quality | Urban fathers<br>who are 18+<br>years with<br>children up to<br>24 years | Assessment of healthy partner relationship behavior at GWA Project enrollment | Participants who complete primary and support services will report healthier partner relationship behavior one year after GWA | Confirmatory |

| Improvement | Project |
|---------------|-------------|
| (CQI) Process | enrollment. |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 2. BACKGROUND

For each <u>outcome research question listed in 1.1</u>, whether descriptive or impact design, briefly summarize the previous literature or existing research that informs the stated research question and how the evaluation will expand the evidence base. Explain why the research questions are of specific interest to the program and/or community. Only a short summary paragraph description is needed below. Additional documentation, such as a literature review, may be appended to this document.

| Research<br>Question<br><i>Topic</i> | Existing Research | Contribution to the Evidence Base | Interest to the Program and/or Community |
|---|---|---|---|
| R1 and<br>R2 | Low-income fathers can lack the <b>parenting skills</b> to fulfill their familial obligations as a parent to promote healthy family relationships. | Determine the extent to which the delivery of GWA Project services enhance the parenting skills of low-income fathers. | Inform practitioners about whether GWA Project design promotes healthy family relationships by improving parent behavior. |
| R3 | Low-income fathers can lack the <b>co-parenting skills</b> to fulfill their familial obligations as a parent to promote healthy family relationships. | Determine the extent to which the delivery of GWA Project services enhance the co-parenting skills of low-income fathers. | Inform practitioners about whether GWA Project design promotes healthy family relationships by improving co-parent behavior. |
| R4 | Low-income fathers can lack the <b>relationship skills</b> to fulfill their obligations as a <b>partner</b> to promote healthy family relationships. | Determine the extent to which the delivery of GWA Project services enhance the partner relationship skills of low-income fathers. | Inform practitioners<br>about whether GWA<br>Project design<br>promotes healthy family<br>relationships by<br>improving partner<br>relationship behavior. |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 3. HYPOTHESES

For each specified research question, state the hypothesized result(s) and briefly describe why these results are anticipated.

| Research Question | Hypothesized Result |
|---|---|
| R1 | Participants will report <b>healthier parenting behavior</b> after the complete <i>primary</i> services and employment support services in the GWA Project. |
| R2 | Participants will report <b>healthier parenting attitudes</b> after the complete <i>primary services</i> and <i>employment support services</i> in the GWA Project. |
| R3 | Participants will report <b>healthier co-parenting behavior</b> after the complete <i>primary services</i> and <i>employment support services</i> in the GWA Project. |
| R4 | Participants will report <b>healthier partner relationship behavior</b> after the complete <i>primary services</i> and <i>employment support services</i> in the GWA Project. |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 4. RESEARCH DESIGN

For each research question, briefly describe why the research design proposed will answer each research question(s). State whether the proposed evaluation is a descriptive or impact evaluation and justify why the proposed research design is best suited to answer the research question(s).

| Research<br>Question | Design | Justification |
|---|---|---|
| R1 | Pre to post outcomes assessment of GWA participation for healthy parenting behavior. | Healthy change reported by participants in their parenting behavior from pre to post estimates the maximum amount of benefit that can be attributed to GWA services in the absence of a counterfactual. |
| R2 | Pre to post outcomes assessment of GWA participation for healthy parenting attitudes. | Healthy change reported by participants in their parenting attitudes from pre to post estimates the maximum amount of benefit that can be attributed to GWA services in the absence of a counterfactual. |
| R3 | Pre to post outcomes assessment of GWA participation for healthy co-parenting behavior. | <b>Healthy</b> change reported by participants in their <b>co-parenting behavior</b> from pre to post estimates the maximum amount of benefit that |

| | | can be attributed to GWA services in the absence of a counterfactual. |
|---|---|---|
| R4 | Pre to post outcomes assessment of GWA participation for healthy partner relationship behavior. | Healthy change reported by participants in their partner relationship behavior from pre to post estimates the maximum amount of benefit that can be attributed to GWA services in the absence of a counterfactual. |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

#### 5. ONGOING GRANTEE AND LOCAL EVALUATOR COORDINATION

Describe how the grantee and local evaluator collaboratively worked together to identify the research question(s) and research design to ensure its feasibility and relevance. Describe how the grantee and local evaluator will continue to work together throughout the evaluation to proactively address unforeseen challenges as they arise and ensure the rigor and relevance of the evaluation and its findings. Describe how the grantee and local evaluator will coordinate dissemination efforts. Describe how these processes will occur while maintaining the independence of the evaluation.

Fathers Incorporated and the local evaluator, Midwest Evaluation and Research (MER) began the process of collaboration prior to the release of the Funding Opportunity Announcement (FOA) for this project. This included multiple working meetings to discuss the project and the goals that Fathers Incorporated had for the project, with a specific emphasis on what they had learned as a funded OFA grantee over the last two cohort cycles and what they would like to do differently. This included a discussion of enhancements to the program they believed would enhance participant outcomes, and the resource requirements of these enhancements. Several viable and relevant research question options were developed prior to the FOA and when the FOA was released the team had additional meetings to discuss the program that would be proposed to meet the goals and objectives of Fathers Incorporated and OFA and how well the research question alternatives developed in advance worked with this program outline. Using this extended collaborative process, the research questions were designed that were most relevant and feasible.

The basis for ongoing coordination between Fathers Incorporated and MER is regular communication. This will be accomplished by the way of bi-weekly meetings and daily interactions between staff. Fathers Incorporated and MER have established a set of standing calls and meetings which begam in the first quarter of funding. This includes a bi-weekly (every other week) meeting of the CQI team. This is a team that is led by the CQI Data Manager and MER Lead Evaluator will discuss program implementation, data from the nFORM and local evaluation systems and closely examine trends and accomplishments (see CQI section for more detail on these meetings). This team includes Fathers Incorporated organizational and project leadership, the MER Evaluation team, and front-line staff in the form of Case Manager and Facilitator representatives.

In addition to this CQI team, a monthly meeting of program and organization leaders and MER staff will occur the ensure the partnership and coordination is on track and running smoothly. Regular contact allows close coordination. Perhaps the greatest asset to this coordination effort is the CQI Data Manager which is a shared and co-funded staff person that is embedded

with Fathers Incorporated staff and acts as staff for both MER and Fathers Incorporated-bridging the gap between the organizations.

This person will interact with program staff daily while completing the duties of a CQI Data Manager. These meetings and staffed position will continue during the entire project period and will include addressing opportunities for dissemination (shared efforts with project staff) and ensuring the rigor and relevance of the evaluation and its findings.

MER has operated prior RCT evaluations with this exact process, by clearly outlining roles and responsibilities – such as the evaluation team helps identify and illuminate areas of concern or improvement (for the program and the evaluation), but the program staff have responsibility for implementing program improvement and for providing direct services to participants.

Fathers Incorporated and MER share a responsibility for a well-executed project and evaluation, but MER is also an independent and external organization that has high integrity and is not responsible in the outcomes of the program. This allows for a high level of coordination without allowing any co-dependence or for personal interests to influence evaluation findings. This was well demonstrated in MER's last evaluation which found the program enhancements being studied ineffective in improving outcomes.

# 6. LEAD STAFF

Define the roles of lead staff for the evaluation from both organizations below.

| Name | Organization | Role in the Evaluation |
|---|---|---|
| Dr. Matthew Shepherd | Midwest Evaluation and Research | Principal Investigator |
| McKenna LeClear | Midwest Evaluation and Research | Senior Research Consultant |
| Dr. Saloni Sharma | Midwest Evaluation and Research | Evaluation Project Manager |
| Darris McKenzie | Fathers Incorporated | CQI Data Manager |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

Articulate the experience, skills, and knowledge of the staff for the evaluation (including whether they have conducted similar studies in this field), as well as their ability to coordinate and support planning, implementation, and analysis related to a comprehensive evaluation plan.

Dr. Matthew Shepherd will serve as the Principal Investigator for this grant. As such, he has corporate responsibility for all evaluation activities. Dr. Shepherd has over 25 years' experience in program design and implementation, applied research, program evaluation, policy analysis, and evaluative technical assistance.

McKenna LeClear will serve as the Senior Research Consultant and provide oversight for HMRF evaluation activities as needed. Ms. LeClear has 5 years of evaluation research experience and oversees numerous other HMRF evaluations for MER.

Dr. Saloni Sharma will serve as the Evaluation Project Manager and will lead the effort to conduct a descriptive study and a Continuous Quality Improvement (CQI) process for the grant. Dr. Sharma has over 5 years or experience in Public Policy research prior to her time at MER.

Darris McKenzie will serve as the CQI Data Manager. He possesses the managerial and analytic skills to successfully serve in this position. The CQI Data Manager will work closely with the grantee and community partners on-site to complete data collection and management activities for the descriptive study <u>and</u> a Continuous Quality Improvement (CQI) process.

#### 7. SAMPLE

# 7.1. TARGET POPULATION(S)

For each target population identified in Section 1.2, please describe the target population(s), and explicitly state whether the population(s) differs from those who will be broadly served by the grant. Describe how the target population will be identified. Explicitly state the unit of analysis (e.g., non-residential father, unmarried couple).

| Description of Target Population | How is the population different from those who will be broadly served by the grant? | How will the target population be identified? | Unit of<br>Analysis |
|---|---|---|---|
| Urban fathers age<br>18 years and older<br>with children who<br>are up to 24 years<br>of age | No difference, all program participants will be study participants | The sample will be identified and recruited by the program staff. | Urban fathers |

#### 7.2. METHODS TO PROMOTE SUFFICIENT PROGRAM PARTICIPATION

Please describe methods to promote sufficient program participation in the table below.

# 8. DATA COLLECTION

# **8.1. CONSTRUCTS AND MEASURES**

Clearly articulate the constructs of interest, measures to evaluate those constructs, and specific data collection instruments. Provide any information on the reliability and validity of the data collection instruments. For standardized instruments, you may provide the citation for the instrument.

| Construct | Measure | Instrument | Reliability and Validity (if standardized instrument, you provide a citation for the instrument) |
|---|---|---|---|
| Parenting<br>Attitudes | 7 items:<br>frequency of key<br>attitudes<br>(categories, 5-<br>point scale) | nFORM<br>Community-<br>Based Fathers<br>Survey (A3: a-g) | nFORM |
| Parenting<br>Behavior | 1 item: hours<br>spent w/ children<br>in last 30 days<br>(interval); 1 item:<br>frequency reach<br>out to children<br>(categories, 5<br>point scale); 7<br>items: frequency<br>engage in key<br>behaviors<br>(categories, 5-<br>point scale) | nFORM<br>Community-<br>Based Fathers<br>Survey (A2b,<br>A2c, A5b: b-d, f-i) | nFORM |
| Co-Parenting<br>Behavior | 11 items:<br>frequency of<br>agreement with<br>key co-parenting<br>behaviors<br>(interval, 5-point<br>scale) | nFORM<br>Community-<br>Based Fathers<br>Survey (A13: a-k) | nFORM, OLLE |
| Healthy<br>Partner<br>Behavior | 1 item: feelings of<br>being<br>overwhelmed as<br>parent<br>(categories, 4<br>point scale) | nFORM<br>Community-<br>Based Fathers<br>Survey (B3 –<br>B3a) | nFORM |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

#### 8.2. CONSENT

Describe how and when program applicants will be informed of the study and will have the option of agreeing (i.e., consenting to) or declining to participate in the study.

Fathers Incorporated staff will make initial contact with interested applicants. They will describe the study and answer any questions at that time. If the applicant is interested in the project, he will be invited to an enrollment session where the consent form will be presented. Fathers Incorporated staff will ensure that the applicant understands the consent form, remind them that participation is voluntary, and that they can drop out of the project at any time for any reason without consequences. Informed consent will take place prior to program enrollment and the collection of evaluation data.

#### 8.3. METHODS OF DATA COLLECTION

If the evaluation will collect multiple waves of data, describe the timing of these waves below. When describing follow-up periods, specify whether the follow-up period will be post-baseline, post-random assignment, or post-program completion.

| Wave of Data Collection (e.g., baseline, short-term follow-up, long-term follow-up) | Timing of Data Collection |
|---|---|
| Baseline | Collected Immediately Following informed consent and enrollment – during and orientation session or first workshop. |
| Post-Test | Collected after the completion of core curriculum programing -during the last workshop session – approximately 13 weeks after enrollment. |
| 1 year Follow-up (post-baseline) | Collected approximately one year after program enrollment/ baseline |

For each measure, describe how data will be collected detailing which data collection measures will be collected by which persons, and at what point in the programming or at what follow-up point.

| Measure | Timing of<br>Data<br>Collection<br>(baseline,<br>wave of data<br>collection) | Method of Data Collection | Who Is<br>Responsible<br>for Data<br>Collection? | Administrative Data Only: Will data access require data sharing agreement? |
|---|---|---|---|---|
| On Line Local<br>Evaluation<br>(OLLE)<br>Baseline<br>Survey | Baseline | Participant<br>Self-Entered<br>survey using<br>online data<br>collection<br>program | Data Manager<br>will proctor<br>data collection<br>and assist<br>participants as<br>necessary | No |
| OLLE Post-<br>Test Survey | Post-Test<br>(approx. 13<br>weeks after<br>enrollment) | Participant<br>Self-Entered<br>survey using<br>online data<br>collection<br>program | Data Manager<br>will proctor<br>data collection<br>and assist<br>participants as<br>necessary | No |
| OLLE 1 Year<br>Follow-up<br>Survey | 1 year after<br>enrollment /<br>baseline | Participant Self-Entered survey using online data collection program and link – or – Phone Interview data collection | MER<br>Research<br>Staff/<br>participant<br>tracking team | No |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

# 8.4. ENSURING AND MONITORING DATA COLLECTION

Describe plans for training data collectors and for updating or retraining data collectors about procedures. Detail plans to regularly review data that have been submitted and to assess and swiftly address problems.

This evaluation will utilize both post-program surveys (completed at the completion of core programing) and follow-up surveys collected one year after enrollment / baseline. The methods for these data collections differ. The primary driver for post-program survey completion is high rates of <u>program</u> retention. This data point will be collected during the last workshop session – after (but during the same session of) the completion of the nFORM post-program data collection. As such only those individuals who complete the program and who are at the data collection session will participate in the post-program data collection.

All program staff and evaluation staff will undergo a rigorous set of trainings to prepare for the evaluation. All staff receive an overview and introductory training to present the goals and objectives of the evaluation effort and its importance to the overall project. Next all staff receive training on human subject's protection and are required to pass a certification test on the subject matter. All staff will also receive a detailed training on the details of the evaluation including the evaluation tools, timing and data collection process.

In addition, the data manager and the primary local evaluation staff will undergo a rigorous training process to better understand the context of HMRF research, training on data collection procedures they will be responsible for, and training on the nFORM system and use of nFORM data in a CQI process. MER is creating networks of CQI data managers and Evaluation Project Managers across the 12 projects that we are evaluating so that all staff have access to experienced data managers and evaluation staff who have done this work previously. This training takes the form of weekly training sessions that are currently under way.

Members of the CQI team will also receive specific training on the MER CQI process that has been developed prior to the launch of data collection or program services. As described elsewhere MER is assisting the program staff in implementing a robust CQI process that will focus on retention as one of the primary areas of program improvement and as such we are anticipating relatively modest levels of attrition for this data collection.

On a bi-weekly basis the data manager, the local evaluation staff and MER technical specialists will be responsible for downloading data from the nFORM and MER On-Line Local Evaluation (OLLE) systems for processing and presentation to the CQI team for tracking and monitoring performance measurement outcomes (recruitment, enrollment, dosage, completion, referrals, etc.) so that near real time adjustments can be made to program implementation to ensure compliance with program goals and objectives.

All MER training is currently being recorded and as new staff come on board with projects or project staff turn over (or need refresher training) recorded training material can be shared and accessed with follow-up one on one training with the primary local evaluator and the MER LOB Lead, who has more than 15 years' experience in evaluating HMRF projects.

# 9. IRB/PROTECTION OF HUMAN SUBJECTS

Please describe the process for protection of human subjects, and IRB review and approval of the proposed program and evaluation plans. Name the specific IRB to which you expect to apply.

Because the planned evaluation involves human subjects, FI understands that program implementation requires both IRB approval and participant informed consent. MER has an established relationship with Solutions IRB MER has had several research studies approved by Solutions IRB, and has submitted timely amendments when changes to studies needed to take effect. Solutions IRB, a private commercial Association for the Accreditation of Human Research Protection Programs Inc. (AAHRPP) fully accredited Institutional Review Board, will ensure that this study is approved before any research activities take place.

All submissions are completed online, so turnaround for a new study approval is between 24 to 72 hours, though the full approval process can take approximately one to two weeks depending on the number of questions and requested revisions that the IRB makes. In the IRB application submission, we will include descriptions of project staff, locations of study sites, the funding source, incentives, summary of activities, participant population, recruitment plans, risks and benefits, confidentiality of data, and the informed consent process along with all materials to be used in the study such as participant forms and surveys.

This project will be submitted for IRB approval in early March during the planning period in order to receive official approval to begin enrollment and data collection beginning in April.

Program staff and facilitators will also obtain Human Subjects Training Certification through the IRB to ensure the protection of participants.

### 10.DATA

# 10.1. DATABASES

For each database used to enter data, please describe the database into which data will be entered (i.e., nFORM and/or other databases), including both performance measure data you plan to use in your local evaluation and any additional local evaluation data. Describe the process for data entry (i.e., who will enter the data into the database).

| Database Name | Data Entered | Process for Data Entry |
|---|---|---|
| nFORM | Performance Measurement<br>Data | Entered directly by participants, and by program staff |
| Qualtrics | Local evaluation data,<br>participant outcomes (OLLE<br>survey) | Entered directly by participants, and by MER evaluation staff |

# 10.2. DATA REPORTING AND TRANSFER

For each database provided in the table above, please indicate the ability to export individual-level reports to an Excel or comma-delimited format and whether identifying information is available for linking to data from other sources.

| Database Name | Ability to Export Individual Reports? | What identifying information is available to facilitate linking to other data sources? |
|---|---|---|
| nFORM | Yes | Client ID, name, DOB |
| Qualtrics | Yes | Client ID, name, DOB |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

#### 10.3. CURRENT SECURITY AND CONFIDENTIALITY STANDARDS

For each database provided in Section 11.1, please Indicate the ability to be able to encrypt data access during transit (for example, accessed through an HTTPS connection); be able to encrypt data at rest (that is, when not in transit), have in place a data backup and recovery plan; require all users to have logins and passwords to access the data they are authorized to view; and have current anti- virus software installed to detect and address malware, such as viruses and worms.

| Database Name | Ability to encrypt data during transit? | Ability to encrypt at rest? | Data Backup and Recovery Plan? | Require all users to have logins and passwords? | Current Anti-<br>Virus Software<br>Installed? |
|---|---|---|---|---|---|
| nFORM | Yes | Yes | Yes | Yes | Yes |
| Qualtrics | Yes | Yes | Yes | Yes | Yes |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

| Please describe any plans for study registration with an appropriate registry (e.g., clinicaltrials.gov, socialscienceregistry.org, osf.io, etc.). |
|---|
| This study will be registered with clinicaltrials.gov. |